CLINICAL TRIAL: NCT01607125
Title: Interventional, Randomised, Double-blind, Parallel-group, Placebo-controlled, Exploratory Study Investigating the Effects of [Vortioxetine] Lu AA21004 on Cognition and BOLD fMRI Signals in Subjects Remitted From Depression and Controls
Brief Title: Exploratory Study of the Effects of Vortioxetine (Lu AA21004) on Cognition and Blood Oxygen Level Dependent (BOLD) Functional Magnetic Resonance Imaging (fMRI) Signals in Subjects Remitted From Depression and in Controls
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14137A; 2011-001839-23 (EudraCT Number)
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vortioxetine (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vortioxetine (Lu AA21004) — encapsulated 20 mg tablets, orally, once daily for 13 to 14 days
  Other Names: Brintellix
  Arms: Vortioxetine
Drug: Placebo — capsules, orally, once daily for 13 to 14 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if Vortioxetine 20 mg/day will lead to changes in neural activity (BOLD signal), as measured using fMRI, in brain areas associated with executive functioning and memory during cognitive task performances compared to placebo in subjects remitted from depression and in controls, and to explore if Vortioxetine will lead to improved cognitive performance in the absence of depression.

ELIGIBILITY:
Inclusion Criteria:

All subjects must have:

* a Hamilton Depression Rating Scale (HAM-D17) total score ≤ 7

Subjects remitted from depression must:

* be in remission from recurrent depression having suffered from at least two previous Major Depressive Episodes (MDEs)
* have received prescribed treatment with an antidepressant or a recognised psychotherapy for depression for a previous MDE
* report present subjective cognitive dysfunction
* not have been treated with antidepressants or received other psychotherapy for depression for at least six weeks prior to screening visit

Control group subjects must:

* have no history of MDEs
* have no history of MDEs in a biological parent or other first degree relative as reported by the subject
* not report present subjective cognitive dysfunction
* never have been treated with antidepressants or psychotherapy

Exclusion Criteria:

* The subject is, in the opinion of the investigator, unlikely to comply with the clinical study protocol or is unsuitable for any other reason

Other inclusion and exclusion criteria may apply.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Effect of Vortioxetine on BOLD signal in fMRI of the brain areas associated with executive function (working memory) | Day 1 to Day 13
Effect of Vortioxetine on BOLD signal in fMRI of the brain areas associated with spatial memory | Day 1 to Day 13

SECONDARY OUTCOMES:
Effect of Vortioxetine on cognitive performance (executive function, memory, speed of processing, attention, cognitive flexibility) and emotional processing | Day 1 to Day 13

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- GB001, Headington, United Kingdom